CLINICAL TRIAL: NCT03483571
Title: Preliminary Evaluation of Dynamics of Subclinical Malaria
Brief Title: Dynamics of Subclinical Malaria: Preliminary Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Ministry of Health and Sports, Myanmar (Other Government); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); National Institute of Parasitic Diseases, China CDC (Unknown); Defence Services Medical Research Center, Myanmar (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00091895
Record Dates: First submitted 2018-03-15; First posted 2018-03-30 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Malaria
Keywords: asymptomatic; submicroscopic; PCR
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — dry blood spot collected on filter papers and venous blood frozen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a short longitudinal preliminary study that aims to describe the dynamics of low-density subclinical malaria to support the final study design of a subsequent matched cohort study. The primary objective is to assess the dynamics of subclinical malaria detected by ultrasensitive PCR over a short duration. The results will be used to guide the design of a matched cohort study of subclinical malaria in Myanmar and along its borders with China and Bangladesh

DETAILED DESCRIPTION:
This is a short longitudinal preliminary study that aims to describe the dynamics of low-density subclinical malaria to support the final study design of a subsequent matched cohort study. In this study, a small number of asymptomatic infections detected by ultrasensitive PCR (usPCR) will be followed and tested intensively for three months to measure the temporal dynamics of these infections. A much larger number of uninfected individuals will be followed for just 2-4 weeks (two visits), providing a comparator group for the infected cohort. The validity of our results in a subsequent matched cohort study depends, in part, on our ability to accurately classify infection status using a single usPCR result. In other words, do the investigators have sufficient confidence in the correct classification of malaria infection positive and negative status using usPCR test at the beginning of the study? While there is no gold standard test more sensitive than usPCR, repeated usPCR testing offers a surrogate. Presumably, in a low transmission setting, someone who is truly uninfected on the first testing should remain negative on multiple consecutive tests, but this remains to be confirmed.

The investigators will enroll study participants in up to six study sites, each with >2 villages, towns, unions, refugee camps or plantations, or a single military base. Alternative and additional sites may be added to ensure enough infected cases. The investigators will screen for eligibility (age at least 0.5 year; able & willing to strictly follow study protocol and to provide written informed consent or assent as appropriate) and enroll and consent eligible individuals. Study procedures are based on test results:

* RDT-positive: one-time enrollment for data and venous blood collection; Refer to and ensure appropriate treatment by care providing team; No study-related follow up
* RDT-negative: Collect data and DBS samples; Return to research clinic in 2-4 weeks
* PCR-negative participants: One follow up visit approximately 2-4 weeks after enrollment
* PCR-positive participants: Five follow up visits at approximately 4, 6, 8, 10, and 12 weeks (for those with total 12 weeks follow up) or 2, 3, 4, 5 and 6 weeks (for those with total 6 weeks follow up) after enrollment
* Finger stick blood sampling with be done for RDT and dried blood spot sampling in all participants at each scheduled and unscheduled visit.
* Venous sampling will be done for participants with RDT+ infections detected at times when study staff trained for venous sampling are present. Blood volumes at any time point are limited to 2 mL for children aged < 3 years, 3 mL for age 3-5 years, and 5 mL for older children and adults.
* Estimated duration of study:18 months

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months or older at the time of screening; Written informed consent obtained (from the parent/guardian if the subject is less than 18 years old).

Exclusion Criteria:

Any condition which in the view of the investigator makes participation not in the best interests of the prospective participant. Any condition that would interfere with study participation or pose risks to participants. Those with clinical malaria infection as diagnosed by positive RDT may be invited to return and be re-screened for study eligibility after treatment and resolution of their illness.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sites broadly representative of the range of malaria epidemiologies seen in the region have been identified based on available data on the incidence of clinical malaria and prevalence of subclinical malaria (measured by both standard testing and by usPCR in surveys we have supported). In a staged fashion, initial screening will be undertaken at these sites, starting with the sites in Myanmar, where laboratories proficient in usPCR have been established.
Sampling Method: Probability Sample
Enrollment: 2970 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Proportion of individuals with initially positive usPCR tests that were followed by 1 or more consecutive positive tests on weekly or biweekly testing | 12 weeks
  Proportion of individuals with initially positive usPCR
Proportion of individuals with initially negative usPCR tests that subsequently had at least one usPCR positive test at a second screening 4 weeks later | 4 weeks
  Proportion of individuals with initially negative usPCR tests

SECONDARY OUTCOMES:
Incidence of falciparum malaria infection by RDT | 2 years
  Incidence of falciparum malaria infection by RDT
Incidence of vivax malaria infection by RDT | 2 years
  Incidence of vivax malaria infection by RDT
Incidence of mixed falciparum/vivax malaria infection by RDT | 2 years
  Incidence of mixed falciparum/vivax malaria infection by RDT
Incidence of falciparum malaria infection by usPCR | 2 years
  Incidence of falciparum malaria infection by usPCR
Incidence of vivax malaria infection by usPCR | 2 years
  Incidence of vivax malaria infection by usPCR
Incidence of mixed falciparum/vivax malaria infection by usPCR | 2 years
  Incidence of mixed falciparum/vivax malaria infection by usPCR
Seroreactivity to polymorphic malaria/mosquito proteins | 2 years
  Seroreactivity to polymorphic malaria/mosquito proteins

CONTACTS AND LOCATIONS:
Overall Officials: Christopher V Plowe, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Department of Medical Research, Yangon, Burma

IPD SHARING:
Plan to Share IPD: No
PID will not be shared with other researchers

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT03483571/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT03483571/ICF_001.pdf